CLINICAL TRIAL: NCT01915381
Title: Improving Adherence Healthy Lifestyle on a Smartphone Based on Complementation Adults With Intellectual Disabilities
Brief Title: Improving Adherence Healthy Lifestyle With a Smartphone Application Based on Adults With Intellectual Disabilities
Acronym: APPCOID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaga (Other)
Responsible Party: Principal Investigator, Dr. Antonio I Cuesta-Vargas, PhD, University of Malaga
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: FCCSS
Record Dates: First submitted 2013-07-23; First posted 2013-08-02 (Estimated); Last update posted 2019-09-30 (Actual); Status verified 2017-02

CONDITIONS: Intellectual Disability
Keywords: Intellectual disability; mHealth; App; Physical activity; Adherence
MeSH Terms: conditions — Intellectual Disability; Alzheimer Disease; Motor Activity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control group (Active Comparator): follow up detraining effect of multimodal intervention
  Interventions: Other: multimodal intervention
- application smartphone-based group (Experimental): Smartphone-based application group (SG) sample will have a reminder to do Phisical activity everyday where patients will have to select if they have done or they haven´t done physical activity.
  Interventions: Other: multimodal intervention

INTERVENTIONS:
Other: multimodal intervention — All subjects received a multimodal intervention consist in a multimodal program with an educational approach, where therapist advice about benefits of PA during the exercises, to promote PA with brochure-based decalogue

SUMMARY:
AIM: Improve adherence to physical activity in people with Intellectual disabilities with a Smartphone Application DESIGN: Randomized controlled trial SUBJECTS OF THE STUDY: People with intellectual disabilities in Occupational Center ( ASPROMANIS) INTERVENTION: DATA ANALYSIS: descriptive statistics, measuring central tendency and dispersion of the variables study. Inferential statistics will be made between intervention of key variables and outcome

ELIGIBILITY:
Inclusion Criteria:

* Participants were can write and read to ask scales
* Participant were able to use an Smartphone

Exclusion Criteria:

* Physical illness that prevent physical activity

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2014-07 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
International Physical activity Questionnaire | up to 8 weeks
  CRAIG, C. L., A. L. MARSHALL, M. SJÖSTRÖM, A. E. BAUMAN, M. L. BOOTH, B. E. AINSWORTH, M. PRATT, U. EKELUND, A. YNGVE, J. F. SALLIS, and P. OJA. International Physical Activity Questionnaire: 12-Country Reliability and Validity. Med. Sci. Sports Exerc., Vol. 35, No. 8, pp. 1381-1395, 2003.

SECONDARY OUTCOMES:
Barthel index | baseline; 8; 18 and 28 weeks
Social Support and Self efficacy SS/SE AID | baseline; 8; 18 and 28 weeks
  The Self-Efficacy and Social Support for Activity for persons with Intellectual Disabilities (SE/SS-AID) scales were developed to measure the relationship between self-efficacy, social support, and physical activity participation for those with ID (Peterson et al., 2009).This modified set of SE/SS-AID scales, composed of 23 questions, and was employed in this study. The Self-Efficacy (SE) scale contained six items, with response options of "no, maybe, and yes." Together, the three Social Support (SS) scales included 17 items, which were divided into three subcategories, including six family items, six staff items, and five peers items. The SS scales have response options of ''no, yes - sometimes, and yes - a lot.''
FunFitness | baseline; 8,18 and 28 weeks
  Funfitness is a battery of 13 fitness tests including: the Passive knee extension test, the Calf muscle flexibility test, the Anterior Hip Flexibility test, the Functional shoulder rotation test, the Timed-stand test, the Partial Sit-up test, the Seated push-up, the Grip test, the Single leg stance open and closed eyes, and the 3 minutes walk test. A detailed description of the tests and data regarding reliability is given Cuesta-Vargas et al Res Dev Disabil. 2011 Mar-Apr;32(2):788-94. doi: 10.1016/j.ridd.2010.10.023. Epub 2010 Dec 15.
Internatioanl Physical Activity Questionnaire (IPAQ) | Changes from 8 weeks during follow up 18 and 28 weeks
  CRAIG, C. L., A. L. MARSHALL, M. SJÖSTRÖM, A. E. BAUMAN, M. L. BOOTH, B. E. AINSWORTH, M. PRATT, U. EKELUND, A. YNGVE, J. F. SALLIS, and P. OJA. International Physical Activity Questionnaire: 12-Country Reliability and Validity. Med. Sci. Sports Exerc., Vol. 35, No. 8, pp. 1381-1395, 2003.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio I Cuesta Vargas, PhD, Principal Investigator — University of Malaga
Locations (1):
- Patronato Municipal de deportes de Torremolinos, Torremolinos, Malaga, Spain

REFERENCES:
- [Derived] Perez-Cruzado D, Cuesta-Vargas AI. Improving Adherence Physical Activity with a Smartphone Application Based on Adults with Intellectual Disabilities (APPCOID). BMC Public Health. 2013 Dec 13;13:1173. doi: 10.1186/1471-2458-13-1173. PMID 24330604
- See also: University of Malaga — http://www.uma.es